CLINICAL TRIAL: NCT03344471
Title: Factors Associated With Post-Traumatic Stress Disorder in Patients With After Preterm Delivery
Acronym: PTSD-preterm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PO17133
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Preterm Delivery
Keywords: preterm delivery; PTSD; prematurity; birth; personality
MeSH Terms: conditions — Premature Birth; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- women with PTSD after preterm deliver (Other)
  Interventions: Other: Passation of questionnaires
- women without PTSD after preterm deliver (Other)
  Interventions: Other: Passation of questionnaires

INTERVENTIONS:
Other: Passation of questionnaires — Specific questionnaires (Perinatal PTSD Questionnaire evaluating the Post-Traumatic Stress Disorder) and (NEO-FFI evaluating personality)

SUMMARY:
Each year in France, between 50,000 and 60,000 children are born prematurely (< 37 weeks of amenorrhea). Literature has shown that preterm deliveries can be associated with the development of PTSD (Post-Traumatic Stress Disorder) in mothers. Around ¼ of women suffer from a PTSD after giving birth prematurely. Moreover, studies highlighted the consequences of a PTSD on the child-mother relationship. Beyond the importance of early detection, it could be important to predict factors that make women more likely to develop a PTSD. This study will focus on personal factors (5 dimensions of personality). Our hypothesis is that personality traits are associated with the likeliness of developing a PTSD after a preterm delivery.

DETAILED DESCRIPTION:
PTSD : Post-Traumatic Stress Disorder. This syndrome can be found in people after they experience a traumatic event. Literature has shown that preterm delivery can lead to the development of PTSD in mothers. PTSD is characterized by symptoms such as:

* Re-experiencing the trauma through intrusive distressing recollections of the event, flashbacks, and nightmares.
* Emotional numbness and avoidance of places, people, and activities that are reminders of the trauma.
* Increased arousal such as difficulty sleeping and concentrating, feeling jumpy, and being easily irritated and angered.

Each year in France, between 50,000 and 60,000 children are born prematurely (< 37 weeks of amenorrhea). Literature has shown that preterm deliveries are associated with the development of PTSD (Post-Traumatic Stress Disorder) in mothers. Around ¼ of women suffer from a PTSD after giving birth prematurely. Moreover, studies highlighted the consequences of a PTSD on the child-mother relationship. Beyond the importance of early detection, it could be important to predict factors that make women more likely to develop a PTSD. This study will focus on personal factors (5 dimensions of personality). Our hypothesis is that personality traits are associated with the likeliness of developing a PTSD after a preterm delivery. ) In order to test our hypothesis, we will have two groups: (1) women who gave birth prematurely and developed a PTSD and (2) women who gave birth prematurely and did not develop a PTSD. Mothers will be recruited in the hospital of Reims a month after delivery. If they accept to participate in the study, a face-to-face-1-hour appointment will be scheduled. During this appointment, women of both groups will take a PTSD questionnaire (the PPQ - Perinatal PTSD Questionnaire) as well as a personality test (the NEO-FFI, see outcome measures) to assess 5 dimensions of their personality (Neuroticism, Extraversion, Openness, Agreeability and Conscientiousness). Individual data will also be collected such as the age of the mother, baby's birth weight, severity of prematurity.

Statistical analyzes will be performed to analyze our results. Student t will be used to compare factors associated with PTSD between both groups. Correlation tests (such as Bravais-Pearson) will also be used to highlight links between personality dimensions and the likeliness to develop a PTSD after a preterm delivery.

NB: Although no intervention is planned in this research, every woman getting a positive score in the PPQ will be addressed to the department's psychologist.

ELIGIBILITY:
Inclusion Criteria:

* mothers who have given birth prematurely (<33 weeks of amenorrhea)
* mothers who speak French fluently
* mothers consenting to participate to the study
* mothers enrolled in the national healthcare insurance program
* mothers older than 18 years

Exclusion Criteria:

* mothers with acute or chronic psychotic disorders,
* mothers with alcohol and/or drug abuse or dependence

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-12-14 (Actual)

PRIMARY OUTCOMES:
PPQ (Perinatal PTSD Questionnaire) | Day 0
  The PPQ is widely used to assess symptoms of PTSD after preterm delivery.
NEO-FFI | Day 0
  self-administered questionnaire used to measure 5 dimensions of personality (Neuroticism, Extraversion, Openness, Agreeability and Conscientiousness)

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France